CLINICAL TRIAL: NCT02190799
Title: Anti-MERS-COV Convalescent Plasma Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC13-244
Record Dates: First submitted 2014-06-12; First posted 2014-07-15 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Respiratory Distress Syndrome (& [Hyaline Membrane Disease])
Keywords: Corona Virus; Convalescent plasma; Serology
MeSH Terms: conditions — Respiratory Distress Syndrome; Hyaline Membrane Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Convalescent plasma (Experimental): Enrolled patients will receive 2 units of the convalescent plasma after meeting the eligibility criteria
  Interventions: Biological: Convalescent plasma

INTERVENTIONS:
Biological: Convalescent plasma — Convalescent plasma from patients who recently recovered from MERS-CoV, HCWs who had potential exposure and subjects who are willing to donate plasma and have their blood tested for anti MERS-CoV serology and RT-PCR after obtaining their consent

SUMMARY:
Since the first report of the Middle East Respiratory Syndrome Corona virus (MERS- CoV) in September 2012, more than 800 cases have been reported to the World Health Organization (WHO) with substantial mortality.

DETAILED DESCRIPTION:
World knowledge about this virus is accumulating but data about the clinical presentations of infected patients and common treatments, including ribavirin, interferon and methylprednisolone, lack evidence. Although drugs with anti- coronavirus (CoV) activities have been identified, as yet no anti- MERs- CoV drug has been approved and a vaccine has yet to be developed. Previous reports on other viral infections including SARS have suggested that convalescent plasma or serum is effective where no other treatment is available or in an emergency. A recently completed systematic review and meta-analysis by the University of Nottingham - World Health Organization Collaborating Center indicates that convalescent plasma therapy may be the most promising near-term therapy patients with for MERS- CoV infection. In this study, investigators will study the pharmacokinetics of immunoglobulin in response to convalescent plasma administration in order to inform a much larger study which will investigate the efficacy of convalescent plasma. Plasma will be collected from patients who recently recovered from MERS-CoV, Health Care Workers who had potential exposure and are tested for anti MERS-CoV serology and RT-PCR after obtaining their consent. This convalescent plasma will be stored in the blood bank as per their policies and procedures. Patients with MERS-CoV positive after meeting the eligibility criteria will receive 2 units of convalescent plasma . Clinical data as well as the standard laboratory studies will be collected at baseline, 30 mins after first dose, 30 mins after second dose, day 1, 3, 7, 14, 28 of hospital stay after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 14 years of age
* Inpatients who are MERS-COV positive (by PCR)
* Willingness to have blood, respiratory and urine samples obtained and stored for subsequent analysis.

Exclusion Criteria:

* Clinical evidence (in the judgment of the site investigator) that the etiology of illness is primarily not MERS-CoV in origin.
* History of allergic reaction to blood or plasma products (as judged by the investigator)
* Known IgA deficiency
* Medical conditions in which receipt of 500mL volume may be detrimental to the patient (e.g., decompensated congestive heart failure)
* Females who are pregnant or breast feeding.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Hospital mortality | Death in the Hospital (ICU or ward) before or at 6 months after enrollment
  Hospital mortality will be death in the ICU during the same hospital admission

SECONDARY OUTCOMES:
ICU mortality | Death in the ICU at or after 90 days of enrollment
  Death in the ICU during the same hospital admission.
ICU Length of Stay | Number of days in ICU with an average expected duration of 10 days.
  Number of calendar days between admission and final discharge from ICU.
Duration of Mechanical Ventilation | Number of days of mechanical ventilation with an expected average duration of 8 days
  Number of calendar days between start and final liberation from mechanical ventilation.
Viral load in tracheal aspirate | Serial levels in the first 28 days of enrollment
  viral clearance from all sampled sites by day 3 after administration of CP
Inflammatory markers, | Serial levels in the first 28 days of enrollment
  Epidermal Growth Factor (EGF), Eotaxin, Granulocyte colony-stimulating factor (G-CSF), Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF), Interferon(IFN)-γ, IFN-a2, Interleukin (IL)-10, IL-12(p40), IL-12(p70), IL-13, IL-15, IL-17, IL-1ra, IL-1a, IL-1β, IL-2, IL-3, IL-4, IL-5, IL-6, IL-7, IL-8, Interferon gamma-induced protein (IP)-10, Monocyte Chemotactic Protein (MCP)-1, Macrophage Inflammatory Protein (MIP)-1a, MIP-1β, Tumor Necrosis Factor-α (TNF-a), TNF-β, Vascular Endothelial Growth Factor (VEGF)
Anti-MERS-CoV antibodies | Serial levels in the first 28 days of enrollment
  anti-MERS-CoV antibody level before and after administration of CP.

OTHER OUTCOMES:
Chest X ray | Serial changes in the X ray till day 28
  X ray changes at day 0, 1, 3, 7, 14, 21 and 28

CONTACTS AND LOCATIONS:
Overall Officials: Yaseen M Arabi, MD, Principal Investigator — King Abdullah International Medical Research Center
Locations (1):
- Intensive Care Unit, King Abdulaziz Medical City, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Arabi Y, Balkhy H, Hajeer AH, Bouchama A, Hayden FG, Al-Omari A, Al-Hameed FM, Taha Y, Shindo N, Whitehead J, Merson L, AlJohani S, Al-Khairy K, Carson G, Luke TC, Hensley L, Al-Dawood A, Al-Qahtani S, Modjarrad K, Sadat M, Rohde G, Leport C, Fowler R. Feasibility, safety, clinical, and laboratory effects of convalescent plasma therapy for patients with Middle East respiratory syndrome coronavirus infection: a study protocol. Springerplus. 2015 Nov 19;4:709. doi: 10.1186/s40064-015-1490-9. eCollection 2015. PMID 26618098